CLINICAL TRIAL: NCT04849559
Title: VP-VLY-686-1301: A Single Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of Tradipitant on Satiation, Gastric Volume, Gastric Accommodation and Gastric Emptying in Healthy Volunteers
Brief Title: Effects of Tradipitant on Satiation, Gastric Volume, Gastric Accommodation, and Gastric Emptying in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VP-VLY-686-1301
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2021-04

CONDITIONS: Healthy Volunteer
Keywords: tradipitant; NK-1 antagonist; neurokinin 1 receptor

STUDY DESIGN:
Intervention Model Description: A single center, randomized, double-blind, placebo-controlled study to evaluate the effects of tradipitant on satiation, gastric volume, gastric accommodation and gastric emptying in healthy volunteers
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tradipitant (Experimental): Oral Capsule
  Interventions: Drug: Tradipitant
- Placebo (Placebo Comparator): Oral Capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tradipitant — Tradipitant Capsule
  Arms: Tradipitant
Drug: Placebo — Placebo Capsule
  Arms: Placebo

SUMMARY:
To evaluate the effects of tradipitant relative to placebo on satiation, gastric volume, gastric accommodation, and gastric emptying in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written consent
* Body Mass Index (BMI) of 18-35 kg/m2
* No medical problems or chronic diseases

Exclusion Criteria:

* Diagnosis of gastrointestinal diseases
* Structural or metabolic diseases that affect the GI system
* A positive test for drugs of abuse at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09-24 (Actual); Study Completion 2021-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanda Pharmaceuticals, Study Director — Vanda Pharmaceuticals
Locations (1):
- Vanda Investigational Site, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khanna L, Zheng T, Atieh J, Torres M, Busciglio I, Carlin JL, Xiao M, Harmsen WS, Camilleri M. Clinical trial: a single-centre, randomised, controlled trial of tradipitant on satiation, gastric functions, and serum drug levels in healthy volunteers. Aliment Pharmacol Ther. 2022 Jul;56(2):224-230. doi: 10.1111/apt.17065. Epub 2022 May 29. PMID 35644931

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tradipitant | Placebo
Started | 13 | 14
Completed | 11 | 13
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tradipitant | Placebo | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (9.61) | 34.9 (10.70) | 33.7 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Fasting Gastric Volume as Measured by Single Photon Emission Computed Tomography (SPECT)
Description: Fasting Gastric volume
Time Frame: 9 Days
Population: Completed subjects
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 11 | 13
mL | 178.8 [158.0 to 217.0] | 191.1 [169.2 to 216.9]

2. Primary Outcome: Accommodation Volume as Measured by SPECT
Description: Gastric Accommodation post 300mL Ensure
Time Frame: 9 Days
Population: Completed subjects
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 11 | 13
mL | 423.8 [358.5 to 484.1] | 411.0 [358.3 to 476.3]

3. Primary Outcome: Satiation Expressed as Volume to Fullness as Measured by Satiation Test
Time Frame: 9 Days
Population: Completed subjects
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 11 | 13
mL | 592.5 [474.0 to 829.5] | 711.0 [474.0 to 948.0]

4. Primary Outcome: Gastric Emptying Half-time of Solids as Measured by Scintigraphy
Description: Gastric Emptying Solids, T50%, Min
Time Frame: 9 Days
Population: Completed subjects
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 11 | 13
minutes | 137.0 [106.8 to 145.0] | 134.0 [125.3 to 141.7]

ADVERSE EVENTS:
Time Frame: 9 days
Description: Safety population includes all subjects enrolled. Efficacy data includes all subjects completed.
Arm/Group | Tradipitant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 4/13 | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tradipitant (N=13) | Placebo (N=14)
fatigue (General disorders) | 2 | 1
peripheral swelling (General disorders) | 1 | 0
swelling face (General disorders) | 0 | 1
abdominal pain (General disorders) | 0 | 1
diarrhea (Gastrointestinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
somnolence (Nervous system disorders) | 2 | 1
headache (Nervous system disorders) | 1 | 1
disturbance in attention (Nervous system disorders) | 1 | 0
dizziness postural (Nervous system disorders) | 1 | 0
restless leg syndrome (Nervous system disorders) | 1 | 0
depressed mood (Psychiatric disorders) | 1 | 0
libido decreased (Psychiatric disorders) | 1 | 0
increased appetite (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT04849559/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT04849559/SAP_001.pdf